CLINICAL TRIAL: NCT02722460
Title: Prospective Registry of Cardiopulmonary Arrest Survivors - Surrogate Markers for Prognostication of Outcome After Cardiac Arrest
Brief Title: Resuscitation Registry - Surrogate Markers of Outcome After Cardiac Arrest
Acronym: CPR
Status: Completed | Type: Observational
Sponsor: Matthias Haenggi (Other)
Responsible Party: Sponsor-Investigator, Matthias Haenggi, Attending Physician, Departement of Intensive Care Medicine, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: KEK BE 116/15
Record Dates: First submitted 2016-03-02; First posted 2016-03-30 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to determine surrogate markers for prognostication of unfavorable outcome (death or persistent vegetative state) in cardiopulmonary arrest survivors. These patients are comatose. Conscious patients are unsuitable for prognostication.

DETAILED DESCRIPTION:
The aim of the study is to determine surrogate markers for prognostication of unfavorable outcome (death or persistent vegetative state) in cardiopulmonary arrest survivors. These patients are comatose. Conscious patients are unsuitable for prognostication.

This will be a prospective mono-center survey (Department of Intensive Care Medicine, University Hospital Bern), evaluating the survival and neurological outcome after cardiac arrest. The study will be performed in cooperation with the Department of Neurology and Neuroradiology, University Hospital Bern.

Inclusion: all patients surviving resuscitation after cardiac arrest older than 18 years. Detailed medical and neurological examination including 6-lead continuous EEG, 10/20 EEG and somatosensory evoked potentials, standard blood tests including Neuron-specific Enolase (NSE) and cerebral MRI will be assessed during the first 72 hours after cardiac arrest. Structured telephone interviews to determine outcome parameters (Cerebral Performance Category CPC, modified Ranking Scale mRS) will take place at day 30, after 3 and 12 month.

The results of the registry could identify early comatose patients after cardiac arrest with no chance of a good neurological recovery and regain consciousness to avoid unjustified expectations of relatives and prolonged life-sustaining therapies. A good neurological recovery is defined as a CPC of 1 and 2 or a mRS 0-2. An unfavourable neurological outcome will be defined as persistent vegetative state and death (CPC 4 and 5, mRS 5-6).

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Down time ≤ 20 minutes (down time = time breakdown to start of professional resuscitation)
* Persistent stable circulation without further need of CPR
* Glasgow Coma Scale < 8 after return of spontaneous circulation

Exclusion Criteria:

* Cardiac arrest due to neurological causes (stroke, intracerebral hemorrhage, subarachnoid hemorrhage, SUDEP - sudden unexpected death in epilepsy)
* Cardiac arrest due to unobserved asystole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with in or out of hospital cardiac arrest and a Glasgow Coma Scale below 8 after emergency service arrived who fulfill the inclusion criteria and none of the exclusion criteria will be included in the prospective registry.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-01; Primary Completion 2021-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
incidence of survival | 30 days after CPR
  incidence of patients still alive 30 days after cardiac arrest or patients discharged alive from hospital

SECONDARY OUTCOMES:
incidence of unfavorable outcome after cardiac arrest according to Cerebral Performance Categories Scale | 72 hours after CPR
  incidence of death within the first 72 hours after cardiac arrest and of death or unfavorable outcome according to the Cerebral Performance Categories Scales 4 and 5 (CPC 4 - Coma or vegetative state: any degree of coma without the presence of all brain death criteria. Unawareness, even if appears awake (vegetative state) without interaction with environment; may have spontaneous eye opening and sleep/awake cycles. Cerebral unresponsiveness, CPC 5 - Brain death)
Number of Patient with a low voltage EEG, defined as amplitude below 20 microvolt more than 24 to 72 hours after resuscitation. | up to 72 hours after CPR
Number of patients with a Cut-off Value of Neuron specific enolase >/= 33 ug/l 72 hours after resuscitation | 72 hours after CPR
Number of patient with a burst suppression EEG more than 24 to 72 hours after resuscitation | up to 72 hours after CPR
Number of patients with an isoelectric EEG more than 24 to 72 hours after resuscitation | up to 72 hours after CPR

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Takala, MD, PhD, Study Chair — Director Department of Intensive Care Medicine University Hospital Bern (Inselspital)
Locations (1):
- Department of Intensive Care Medicine University Hospital Bern (Inselspital), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kagi E, Weck A, Iten M, Levis A, Haenggi M. Value of the TTM risk score for early prognostication of comatose patients after out-of-hospital cardiac arrest in a Swiss university hospital. Swiss Med Wkly. 2020 Sep 9;150:w20344. doi: 10.4414/smw.2020.20344. eCollection 2020 Sep 7. PMID 32920792